CLINICAL TRIAL: NCT04640506
Title: Accuracy of Assessing the Gingival Biotype in the Anterior Maxillary Area in Adult Patients, Using Different Measurement Methods.
Brief Title: Accuracy of Assessing the Gingival Biotype in Upper Anterior in Adult Patients, Using Different Methods.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fahd Ayad Hammoodi Al-Janabi, Principal investigator, Cairo University
Other Study IDs: PER -3-3-1
Record Dates: First submitted 2020-09-25; First posted 2020-11-23 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a Diagnostic accuracy study that determining the accuracy of assessing the gingival biotype and some other anatomic parameters,including (crown width / crown length ratio, attached gingival width, labial bone thickness and papilla volume) by different methods :1- probe transparency, 2-transgingival probing, 3-cone beam computed tomography, 4-intraoral digital scanning, 5-extraoral digital scanning

DETAILED DESCRIPTION:
* Patients will be recruited in periodontic department faculty of dentistry Cairo university.
* Patients who already need esthetic rehabilitation treatment (implant placement, restorative treatments, periodontal therapy, and root coverage) on anterior maxilla and this treatment needs to investigate the gingival biotype.
* Medical history will be taken.
* Oral examination will be done.
* Full mouth periodontal examination and charting will be done for each patient.
* The investigation will be explained to the patient.
* All the investigations will be carried out by one investigator.
* Dental patients will be received to the clinic (for esthetic rehabilitation treatment such as implant placement, restorative treatments, periodontal therapy, and root coverage on anterior maxilla).
* Patients who needs treatment will be investigated the gingival biotype by the five measurement methods (PT, TP, CBCT, IDS and EDS).
* Patients refusing to participate will be reported with the cause of their refusal.
* Conventional clinical examination will be held on a dental unit using the light of the unit, mirror and probe.
* Before the investigation, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be obtained.
* Periodontal status will be evaluated including assessment of gingival index (GI), plaque index (PI), probing pocket depth (PPD) on aesthetic zone in maxillary teeth by using UNC 15 periodontal probe which is 15mm long probe with markings at each millimetre and colour coded at 5th,10th and 15th mm.
* Then an investigator will evaluate the gingival biotype by probing Transparency (PT) as reported by (Kan et al., 2010). The periodontal probe will be softly inserted into the gingival sulcus till it reaches the sound bone on the labial side of the maxil¬lary anterior teeth and it will be parallel to the long axis of the crown. The gingival biotype will be considered as thick if the probe tip is not seen into the tissue and it will be considered as thin if the probe was seen. If the thick en d of the probe was seen into the tissue but the thin end was not, then it will be considered as a moderate biotype.
* The second method of assessment to the gingival biotype will be carried out using CBCT with lip retraction. It is important to note that the patients will not receive additional radiation exposure for the purpose of this investigation and to give us clear details about soft tissue, patients have already underwent CBCT examination as an investigation method for aesthetic rehabilitation treatment.
* Afterwards, gingival biotype assessment will be done by intraoral digital examination (Kim et al., 2016). This is the third method; the investigation of gingival biotype of the anterior maxilla will be done by means of a three-dimensional intraoral scanner. The intraoral scanning data will be acquired in stereolithogra¬phy (STL) format and will be matched with the CBCT data. Three highly radiopaque and relatively fixed positions in the teeth will be chosen as fiducially markers to match the STL files with the CBCT images in accordance with a best-fit algorithm using TRIOS software (3Shape).
* Finally, the fourth method for gingival biotype investigation will be performed by extraoral digital scanning (EDS) of a gypsum cast of the maxillary teeth, then the classic alginate impression of the max-illary arch and cast with dental stone will be made, gyp¬sum cast will be scanned using a three-dimen-sional scanner, and the STL data will be matched with the CBCT image according to a best-fit algorithm as in intraoral method.
* Assessment of some anatomic parameters (crown width/crown length ratio, attached gingival width, labial bone thickness and papilla volume) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Patients whose age is between 18 to 40 years old.
2. Health teeth only will be included.
3. Patients who already need esthetic rehabilitation treatment (implant placement, restorative treatments, periodontal therapy, and root coverage) on anterior maxilla and this treatment needs to investigate the gingival biotype.
4. An un-inflamed periodontal condition with a periodontal probing depth of no more than 3 mm, a bleeding index of < 2, and no gingival recession on maxillary anterior teeth.
5. Provide informed consent.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Restoration or crowns in the maxillary anterior dentition.
3. Malocclusion.
4. Use of any medication affecting the soft tissue.
5. Cigarette smoking.
6. Individuals with chronic systemic diseases such as diabetes, endocrine and haematological pathologies.
7. Patients having problem in opening their mouth or undergoing inter-maxillary fixation where oral examination will not be possible.
8. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
9. Patients with congenital disorders or craniofacial anomalies such as cleft lip and palate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult Egyptian dental patients receiving esthetic rehabilitation treatment (implant placement, restorative treatments, periodontal therapy, and root cov¬erage) on anterior maxilla at faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
gingival biotype assessment by different methods. | the outcome measure will be assessed and for which data will be reported up to 24 weeks"
  will be assess by different methods measurement
  1. probe transparency (PT)
  2. transgingival probing (TP) , 3-cone-beam computed tomography (CBCT)
  4-intraoral digital scanning (IDS) 5-extraoral digital scanning (EDS)
  I will be measured according to De Rouck et al. :
  * less than 1 mm thin-scalloped biotype'' (cluster A1): ''slender teeth, a narrow zone of keratinized tissue and a highly scalloped gingival margin
  * more than 1 mm 'thick-flat biotype'' (cluster B): A clear thick gingiva was found in about two-thirds quadratic teeth, a broad zone of keratinized tissue and a flat gingival margin
  * more than 1 mm (cluster A2): a clear thick gingiva with slender teeth, a narrow zone of keratinized tissue and a high gingival scallop

CONTACTS AND LOCATIONS:
Locations (1):
- Fahd Ayad hammoodi Al-janabi, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No